CLINICAL TRIAL: NCT02153190
Title: Assessment of Hybrid Use of an Artificial Pancreas in a Home Setting for Two Months in Patients With Type 1 Diabetes
Brief Title: Hybrid Artificial Pancreas in Home Setting
Acronym: AP Hybrid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8628 4
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Type 1 Diabetes Mellitus; Treatement by Insulin Pump
Keywords: Type 1 Diabetes,; T1DM,; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HYBRID-OPEN (Experimental): Patients are randomized on the schedule; hybrid period and after open period. During the HYBRID Period, the patient will use the AP model when at home, from dinner to wake-up time whereas the patient will self manage glucose control with insulin pump and CGM for the rest of the day.
  During the control period called OPEN Period, patient self management of diabetes by insulin pump and CGM will be done at all times. Overall, an increase of time spent in range when using artificial pancreas in the hybrid period should be observed with a reduction of both hypo and hyperglycemia episodes.
  Interventions: Device: HYBRID; Device: OPEN
- OPEN-HYBRID (Experimental): Patients are randomized on the schedule: open period and after hybrid period. During the control period called OPEN Period, patient self management of diabetes by insulin pump and CGM will be done at all times.
  During the HYBRID Period, the patient will use the AP model when at home, from dinner to wake-up time whereas the patient will self manage glucose control with insulin pump and CGM for the rest of the day. Overall, an increase of time spent in range when using artificial pancreas in the hybrid period should be observed with a reduction of both hypo and hyperglycemia episodes.
  Interventions: Device: HYBRID; Device: OPEN

INTERVENTIONS:
Device: HYBRID — During the HYBRID Period, the patient will use the AP model when at home, from dinner to wake-up time whereas the patient will self manage glucose control with insulin pump and CGM for the rest of the day.
Device: OPEN — During the control period called OPEN Period, patient self management of diabetes by insulin pump and CGM will be done at all times.

SUMMARY:
The primary purpose of this study is the evaluate an Artificial Pancreas during 2 months in home setting in Type 1 Diabetic patients

DETAILED DESCRIPTION:
During this study, we propose to assess an Artificial Pancreas in a group of Type 1 diabetic patients who will participate in two study periods of two-month duration with an insulin pump and a Continuous Glucose Monitoring (CGM) device. During one of these periods, called HYBRID Period, the patient will use the AP model when at home, from dinner to wake-up time whereas the patient will self manage glucose control with insulin pump and CGM for the rest of the day. During the control period called OPEN Period, patient self management of diabetes by insulin pump and CGM will be done at all times. Overall, an increase of time spent in range when using artificial pancreas in the hybrid period should be observed with a reduction of both hypo and hyperglycemia episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 et < 70 years old
2. Having diabetes according to WHO criteria for at least 6 months, and Type 1 diabetes according to ADA criteria
3. Under basal-bolus insulin therapy using an external insulin pump for at least 3 months
4. BMI < 35 kg/m²
5. Willing to wear a CGM device for the whole duration of the study, except during washout period, combined with the DiAs platform during the evening and night-time for 2 months
6. Trained in carbohydrate counting
7. HbA1c > 7.5 % and < 10%
8. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, stability on the medication for at least 1 month prior to study inclusion
9. Willing to undergo all study procedures
10. Informed consent signed

Exclusion criteria:

1. Pregnancy or breast feeding, or intention to be pregnant during the study duration
2. Use of a medication that significantly impacts glucose metabolism, e.g. steroids
3. Uncontrolled hypertension with resting blood pressure over 140/90 mmHg
4. Patient plans to go abroad during the trial period
5. Patient is expected to be out-of-home in the evening and during night time (e.g. shift-workers, etc.) more than 25% of a study period
6. Patient does not hold any nearby party for assistance if needed
7. Patient with severe hypoglycemia including coma, mental confusion and/or convulsions requesting IV glucose injection or glucagon injection during the last year.
8. Presence of any malignant disease, unless considered as cured for more than 10 years
9. History of acute cardiovascular event during the prior year
10. History of diabetic keto-acidosis during the prior 6 months
11. Renal insufficiency with creatinin > 150 μmol/L
12. Impairment of liver status estimated from ASAT/ALAT plasma levels > 2x upper limits of normal values
13. Impaired cognitive or psychological abilities which may result in defective adherence to study conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percent time spent in target range (3.9-10.0 mmol/L or 70-180 mg/dL) during each study period | during 2 months-hybrid period and during 2 months-open period

SECONDARY OUTCOMES:
Low Blood Glucose Index (LBGI) | for each period of 2 month (hybrid period and open period)

CONTACTS AND LOCATIONS:
Overall Officials: Eric ER RENARD, MD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- CHU Montpellier, Montpellier, France
- University of Padova, Padua, Italy
- University of Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Renard E, Farret A, Kropff J, Bruttomesso D, Messori M, Place J, Visentin R, Calore R, Toffanin C, Di Palma F, Lanzola G, Magni P, Boscari F, Galasso S, Avogaro A, Keith-Hynes P, Kovatchev B, Del Favero S, Cobelli C, Magni L, DeVries JH; AP@home Consortium. Day-and-Night Closed-Loop Glucose Control in Patients With Type 1 Diabetes Under Free-Living Conditions: Results of a Single-Arm 1-Month Experience Compared With a Previously Reported Feasibility Study of Evening and Night at Home. Diabetes Care. 2016 Jul;39(7):1151-60. doi: 10.2337/dc16-0008. Epub 2016 May 5. PMID 27208331
- [Derived] Kropff J, Del Favero S, Place J, Toffanin C, Visentin R, Monaro M, Messori M, Di Palma F, Lanzola G, Farret A, Boscari F, Galasso S, Magni P, Avogaro A, Keith-Hynes P, Kovatchev BP, Bruttomesso D, Cobelli C, DeVries JH, Renard E, Magni L; AP@home consortium. 2 month evening and night closed-loop glucose control in patients with type 1 diabetes under free-living conditions: a randomised crossover trial. Lancet Diabetes Endocrinol. 2015 Dec;3(12):939-47. doi: 10.1016/S2213-8587(15)00335-6. Epub 2015 Sep 30. PMID 26432775